CLINICAL TRIAL: NCT02612194
Title: LCI-GU-URO-CRI-001: A Phase II Study of Crizotinib in Patients With c-MET or RON-Positive Metastatic Urothelial Cancer
Brief Title: LCI-GU-URO-CRI-001: Crizotinib in Patients With c-MET or RON-Positive Metastatic Urothelial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed to accrual due to low accrual numbers.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI-GU-URO-CRI-001
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-05

CONDITIONS: Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): c-MET high (> 50%), RON null (0-9%)
  Interventions: Drug: Crizotinib
- Cohort 2 (Experimental): c-MET + (10-100%), RON + (10-100%)
  Interventions: Drug: Crizotinib
- Cohort 3 (Experimental): c-MET null (0-9%), RON + (10-100%)
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Crizotinib was administered orally at 250mg twice daily
  Other Names: Xalkori

SUMMARY:
This is a single arm two-stage phase II study with crizotinib (Xalkori®) in the treatment of subjects with metastatic urothelial cancer of the bladder, upper (ureter or renal pelvis) or lower (urethra) urinary tracts. The purpose of this study is to see if this experimental drug has a potential benefit in subjects with stage 4 urothelial cancer.

This study tests crizotinib used alone in subjects with urothelial cancer, previously treated with chemotherapy, and whose tumors have certain proteins. Proteins are complex natural substances essential to the structure and function of all living cells. These proteins, c-MET or RON, may trigger molecular pathways that are involved in the growth and spread of bladder or upper urinary tract cancer. Crizotinib is a drug taken by mouth that blocks these pathways. Early laboratory research suggests that crizotinib may benefit patients with urothelial and other cancers with these molecular pathways.

DETAILED DESCRIPTION:
This is a single arm two-stage phase II study designed to evaluate the objective response rate in subjects with metastatic urothelial cancer demonstrating c-MET or RON overexpression who have received prior therapy with a cisplatin or carboplatin containing regimen.

Subjects will be recruited at Levine Cancer Institute (LCI) and other participating sites.

Immunohistochemistry will be utilized to define tumor sample c-MET and RON protein expression patterns for assignment into molecular cohorts as described in section 12.1.

In the first stage of this study, subjects will be enrolled in parallel to three molecularly defined cohorts as follows:

1. c-MET high (>50%), RON null (0-9%) (n = 14 subjects)
2. c-MET-positive (10-100%), RON-positive (10-100%) (n = 7 subjects)
3. c-MET null (0-9%), RON-positive (10-100%) (n = 7 subjects)

All enrolled subjects will continue with study treatment until criteria for treatment discontinuation has been met.

If Stage 1 response criteria are met in a cohort, the cohort may be considered for expansion, and additional subjects (16 in Cohort 1 or 25 in Cohorts 2 or 3) may then be enrolled into that cohort in Stage 2. An expansion cohort will be defined by the Sponsor- Investigator following review of all available trial data which will be conducted after the first Stage 1 cohort has completed accrual and at least every six months thereafter until all Stage 1 cohorts have completed accrual.

If more than one cohort meets Stage 1 response criteria (2 responses out of 14 subjects for Cohort 1 or 1 response out of 7 subjects for each of Cohorts 2 and 3), then the cohort showing the highest response rate will be given highest consideration for expansion.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria:

1. Histologically confirmed stage IV urothelial carcinoma of the bladder, upper urinary tract or urethra.
2. Prior treatment for metastatic disease with at least one cisplatin or carboplatin-based multi-agent chemotherapeutic regimen. Prior immunotherapy with anti-PD-L1 or anti-PD1 agents is allowed.

   o Chemotherapy received peri-operatively for non-metastatic bladder cancer will be considered a prior regimen if less than 24 months have elapsed since treatment.
3. Measurable disease per RECIST 1.1. See Section 10 for the evaluation of measurable disease.
4. Tissue Pre-screen: Archived tissue must have been obtained within 60 months of subject signing tissue pre-screen consent. Biopsy accessible disease if adequate archival tissue does not exist for molecular characterization.

   Treatment: Available tumor specimen C-MET/RON expression results that meet the criteria for one of the three molecularly defined cohorts per Section 4.2
5. Age ≥ 18 years
6. ECOG performance status ≤ 2
7. Adequate liver function: AST and ALT ≤ 2x upper limit of normal, bilirubin ≤ 1.5x upper limit of normal
8. Adequate bone marrow function: Platelets ≥ 100,000 cells/mm3, hemoglobin > 8.0 g/dL and ANC ≥ 1,500 cells/mm3
9. Adequate renal function with a creatinine clearance (based on Cockgroft-Gault formula) ≥ 45 mL/min
10. Ability to understand and the willingness to sign a written informed consent document
11. Able to swallow oral medication

Exclusion Criteria

Subjects must not meet any of the following criteria

1. Currently receiving any other investigational agents, a prior c-MET inhibitor, or crizotinib
2. Pregnant or breast feeding, because crizotinib can cause fetal harm
3. Uncontrolled and current illness including, but no limited to:

   * Ongoing or active infection
   * Symptomatic congestive heart failure
   * Unstable angina pectoris
   * Cardiac arrhythmia, or
   * Psychiatric illness/social situations that would limit compliance with study requirements
4. Presence of any of the following within the previous 3 months of treatment consent:

   * Myocardial infarction
   * Severe/unstable angina
   * Coronary/peripheral artery bypass graft
   * Congestive heart failure, or
   * Cerebrovascular accident including transient ischemia attack
5. History of active malignancy other than urothelial carcinoma within the prior 12 months of the date of treatment consent (except non-melanoma skin cancer or localized, treated prostate cancer)
6. Prolonged QT interval (QTc > 480 msec), symptomatic bradycardia, ongoing cardiac dysrhythmias of CTCAE version 4.0 grade 2 ≥ or uncontrolled atrial fibrillation of any grade
7. Pulmonary disorder requiring supplemental oxygen or history of pulmonary fibrosis. Sleep apnea considered to be a sleep disorder (and not a pulmonary disorder) by the investigator will be allowed.
8. Subjects receiving any medications or substances that are strong inhibitors or inducers of CYP3A are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated list such as http://medicine.iupui.edu/clinpharm/ddis/table/aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the subject will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the subject is considering a new over-the-counter medicine or herbal product.

   * Medical condition requiring the use of strong CPY3A inhibitors, including but not limited to atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, suboxone, telithromycin, troleandomycin, and voriconazole.
   * Use of grapefruit or grapefruit juice, which are considered strong CYP3A inhibitors.
   * Medical condition requiring the use of strong CYP3A inducers, including but not limited to carbamazepine, efavirenz, modafinil, nevirapine, oxcarbazepine, phenobarbital, phenytoin, pioglitazone, rifabutin, rifampin, St. John's Wort, and troglitazone.
9. Receiving any medications that are CYP3A substrates with a narrow therapeutic range (alfentanil, cyclosporine, dihydroergotamine, fentanyl, pimozide, quinidine, sirolimus and tacrolimus)
10. Subjects may be screened for study participation though may not begin study treatment:

    * Within 4 weeks of major surgery
    * Within 2 weeks of prior systemic therapy
    * Within 2 weeks of prior non-palliative radiotherapy
    * Within 48 hours of completion of palliative radiotherapy (≤ 10 fractions)
    * Until recovery of adverse events due to prior therapies to ≤ 1 (except alopecia)
11. Presence of untreated brain metastases or ≤ 6 months from prior treatment (from the time of enrollment), active neurologic symptoms or the use of prohibited medications in subjects with a history of brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Earle Burgess, MD, Principal Investigator — Atrium Health (formerly Carolinas HealthCare System)
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: c-MET high (> 50%), RON null (0-9%)
  Crizotinib: All arms will receive crizotinib.
- Cohort 2: c-MET + (10-100%), RON + (10-100%)
  Crizotinib was administered orally at 250 mg twice daily.
- Cohort 3: c-MET null (0-9%), RON + (10-100%)
  Crizotinib was administered orally at 250 mg twice daily.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 6 | 0 | 2
Completed | 0 | 0 | 0
Not Completed | 6 | 0 | 2
Not completed — Death | 5 | 0 | 2
Not completed — Early Study Termination | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Note, there were no subjects enrolled to cohort 2 as no subjects were enrolled who were c-MET + and RON+. Therefore, no baseline results are available for Cohort 2.
Groups:
- Cohort 2: c-MET + (10-100%), RON + (10-100%)
  Crizotinib: All arms will receive crizotinib.
- Cohort 3: c-MET null (0-9%), RON + (10-100%)
  Crizotinib: All arms will receive crizotinib.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 6 | 0 | 2 | 8
Age, Continuous [Median (Full Range); unit: years] | 60 [53 to 77] |  | 71.5 [64 to 79] | 62 [53 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 0 | 2
  Male | 4 |  | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0 | 0
  Not Hispanic or Latino | 6 |  | 2 | 8
  Unknown or Not Reported | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 1 |  | 0 | 1
  White | 5 |  | 2 | 7
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 |  | 2 | 8
Primary Tumor Site [Count of Participants; unit: Participants]
  Bladder | 5 |  | 1 | 6
  Other | 1 |  | 1 | 2
ECOG at Baseline [Count of Participants; unit: Participants] — Measure Description: ECOG Scale of Performance Status, developed by the Eastern Cooperative Oncology Group, where 0 indicates subject is fully active, able to carry on all pre-disease performance without restriction and where 1 indicates subject is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    0 | 4 |  | 0 | 4
    1 | 2 |  | 2 | 4
c-MET Expression, % [Count of Participants; unit: Participants] — c-MET protein expression was assessed by immunohistochemistray as percent of tumor cells staining positive.
  Participants
    0% | 0 |  | 1 | 1
    1 - 9% | 0 |  | 1 | 1
    51 - 75% | 2 |  | 0 | 2
    >75% | 4 |  | 0 | 4
RON Expression, % [Count of Participants; unit: Participants] — RON protein expression was assessed by immunohistochemistray as percent of tumor cells staining positive.
  Participants
    0% | 2 |  | 0 | 2
    1 - 9% | 4 |  | 0 | 4
    >75% | 0 |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Overall response will be determined as the best treatment response for each patient as a binary variable indicating whether or not the patient achieved a Complete Response (CR) or Partial Response (PR) as determined by RECIST v1.1 criteria. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1):Complete Response (CR) is the disappearance of all lesions (target and non target); Partial Response (PR) is at least 30% decrease in the sum of the diameters of target lesions from baseline and no new lesions or unequivocal progression in non target lesions from baseline; Stable Disease (SD) is neither sufficient shrinkage in target lesions to qualify for PR (less than 30% decrease) nor sufficient increase in target lesions (versus smallest sum of diameters) to qualify for PD (less than 20% increase), with no new lesions or unequivocal progression in non target lesions from baseline. For the purposes of response determination, confirmatory scan for CR and PR is required.
Time Frame: From enrollment to best response while on crizotinib; Subjects remained on treatment until disease progression or death or unacceptable toxicity (subjects were on treatment for an average of 6 weeks)
Population: Study was designed to evaluate objective response rate overall for all enrolled subjects and not separately by molecular cohorts. Efficacy analyses were conducted on the population of subjects who began crizotinib treatment. Analysis of overall response rate was conducted on those patients in the efficacy population with measurable disease present at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Total Enrolled Study Cohort: This group contains all subjects enrolled on the study, who received crizotinib, pooling the subjects in the three molecularly defined cohorts.
Arm/Group | Total Enrolled Study Cohort
Number analyzed (Participants) | 8
Participants | 0
Statistical Analysis 1: Comparison: Total Enrolled Study Cohort; Test type: Other — Estimation only; Overall Response Rate = 0, 95% CI 2-sided [0.000 to 0.369] — Confidence interval estimated using the Clopper Pearson method

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the duration from enrollment date to the date of death from any cause. Subjects who were alive or lost to follow-up at the time of the analysis were censored at the last known date they were alive.
Time Frame: From date of treatment start to date of death, or censored as described above; assessed for approximately 2 years.
Population: Study was designed to evaluate outcomes overall for all enrolled subjects and not separately by molecular cohorts. Efficacy analyses were conducted on the population of subjects who began crizotinib treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Total Enrolled Study Cohort
Number analyzed (Participants) | 8
months | 3.1 [0.2 to 6.1]
Statistical Analysis 1: Comparison: Total Enrolled Study Cohort; Test type: Other — Estimation only; Median = 3.1, 95% CI 2-sided [0.2 to 6.1] — The Kaplan Meier method was used to estimate the median OS (in months) for the population. The Greenwood method was used to estimate the confidence limits of the median overall survival

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as duration of time from enrollment to the study to time of progression or death. Disease progression (PD) can be objectively determined as per RECIST v1.1 (Response Evaluation Criteria in Solid Tumors, where PD is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in non-target lesion, or the appearance of new lesions) or progression can be subjective as determined by the investigator. Evidence for subjective progressions must be documented in medical records. For surviving subjects who do not have documented PD, PFS will be censored at last radiologic assessment. For subjects who receive subsequent anti-cancer therapy prior to documented PD, PFS will be censored at last radiologic assessment prior to commencement of subsequent therapy. Subjects who experience a PFS event following an interval equal to two or more scheduled assessments will be censored at date of last assessment prior to first missed assessment.
Time Frame: From date of treatment start to date of progression or death, or censored as described above; assessed for approximately 2 years.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Total Enrolled Study Cohort
Number analyzed (Participants) | 8
months | 1.5 [0.2 to 1.8]
Statistical Analysis 1: Comparison: Total Enrolled Study Cohort; Test type: Other — Estimation only; Median = 1.5, 95% CI 2-sided [0.2 to 1.8] — The Kaplan Meier method was used to estimate the median PFS (in months) for the population. The Greenwood method was used to estimate the confidence limits of the median progression free survival

ADVERSE EVENTS:
Time Frame: Baseline, during treatment, and through 30 days after last dose. Duration of treatment was the time from treatment start until evidence of progressive disease, unacceptable toxicity, Investigator discretion, or consent withdrawal.
Description: Note, as there were no subjects enrolled in Cohort 2, the number of participants at risk for All-Cause Mortality, Serious Adverse Events, and Adverse Events in Cohort 2 is zero.
Groups:
- Total: Pooled Cohorts 1, 2, and 3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
All-Cause Mortality (participants affected / at risk) | 5/6 | 0/0 | 2/2 | 7/8
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/0 | 2/2 | 4/8
Other Adverse Events (participants affected / at risk) | 5/6 | 0/0 | 2/2 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=0) | Cohort 3 (N=2) | Total (N=8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Fever (General disorders) | 1 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Pain (General disorders) | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=0) | Cohort 3 (N=2) | Total (N=8)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Bloating (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 1 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Creatinine increased (Investigations) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Edema limbs (General disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Eye disorders - Other (Eye disorders) | 1 | 0 | 0 | 1 — Photopsia
Fatigue (General disorders) | 3 | 0 | 2 | 5
Fever (General disorders) | 1 | 0 | 0 | 1
Flashing lights (Eye disorders) | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Floaters (Eye disorders) | 2 | 0 | 0 | 2
Gait disturbance (General disorders) | 0 | 0 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Photophobia (Eye disorders) | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1
Radiculitis (Nervous system disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT02612194/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT02612194/ICF_001.pdf